CLINICAL TRIAL: NCT04507711
Title: The Effect of a Palonosetron on Blood Coagulation: In Vitro, Volunteer Study Using Thromboelastography
Brief Title: Palonosetron and Blood Coagulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B-2002/631-304
Record Dates: First submitted 2020-07-31; First posted 2020-08-11 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 ng/ml (Experimental): Blood specimen which was added of 0 ul of palonosetron
  Interventions: Drug: 0 ul of palonosetron
- 25 ng/ml (Experimental): Blood specimen which was added of 1 ul of palonosetron
  Interventions: Drug: 1 ul of palonosetron
- 250 ng/ml (Experimental): Blood specimen which was added of 10 ul of palonosetron
  Interventions: Drug: 10 ul of palonosetron
- 2500 ng/ml (Experimental): Blood specimen which was added of 100 ul of palonosetron
  Interventions: Drug: 100 ul of palonosetron

INTERVENTIONS:
Drug: 0 ul of palonosetron — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (0 ul) using palonosetron
  Arms: 0 ng/ml
Drug: 1 ul of palonosetron — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (1 ul) using palonosetron
  Arms: 25 ng/ml
Drug: 10 ul of palonosetron — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (10 ul) using palonosetron
  Arms: 250 ng/ml
Drug: 100 ul of palonosetron — Venous blood is taken from 11 healthy volunteers and divided into four specimen bottles, which were added with different doses (100 ul) using palonosetron
  Arms: 2500 ng/ml

SUMMARY:
Palonosetron may alter whole blood coagulation. However, little is known about the dose-response relationships according to the blood concentration of palonosetron. The investigators therefore will perform the present study to measure the effect of palonosetron levels using thromboelastography.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age: 20 to 65 years
* Body weight > 50 kg
* Volunteers who provided informed consent

Exclusion Criteria:

* Hematologic disease
* Anticoagulant medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Citrated Functional Fibrinogen | During the thromboelastography analysis/ an average of 1 hour
  Provides clot strength based on fibrinogen contribution

SECONDARY OUTCOMES:
Citrated Kaolin | During the thromboelastography analysis/ an average of 1 hour
  Normal thromboelastography
Citrated Kaolin Heparinase | During the thromboelastography analysis/ an average of 1 hour
  To assess the effect of heparin
Citrated Rapid Thromboelastography | During the thromboelastography analysis/ an average of 1 hour
  A quicker assessment of clot strength, without assessment of clot initiation
Heparinized Kaloin Heprinase | During the thromboelastography analysis/ an average of 1 hour
  To measure the platelet function
Activator F | During the thromboelastography analysis/ an average of 1 hour
  To elimitate the platelt function
Adenosine diphosphate | During the thromboelastography analysis/ an average of 1 hour
  To measure the drug effect
Arachidonic acid | During the thromboelastography analysis/ an average of 1 hour
  To measure the drug effect

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea